CLINICAL TRIAL: NCT05096598
Title: A First-in-human, Randomised, Single Ascending Dose Trial Assessing Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ZP8396 Administered to Healthy Subjects
Brief Title: A First-in-human Study Looking at the Safety of ZP8396 and How it Works in the Body of Healthy Trial Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP8396-21037; 2021-001712-28 (EudraCT Number); U1111-1267-1489 (Other: WHO)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Overweight; Healthy Volunteers
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: First human dose trial. A single-centre, placebo-controlled, double-blind (within cohorts), randomised single dose trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZP8396 (Experimental): Up to 10 single dose cohorts are planned with 8 subjects in each; 6 participants in each cohort will receive active treatment.
  Interventions: Drug: ZP8396
- Placebo (ZP8396) (Placebo Comparator): In each of the 10 single dose cohorts, 2 subjects will receive placebo.
  Interventions: Drug: Placebo (ZP8396)

INTERVENTIONS:
Drug: ZP8396 — Participants will receive 1 single dose of ZP8396 given subcutaneously (s.c., under the skin) or intravenously (i.v., in a vein of the arm). Dose level will depend on the cohort.
  Arms: ZP8396
Drug: Placebo (ZP8396) — Participants will receive 1 single dose of placebo given subcutaneously (s.c., under the skin) or intravenously (i.v., in a vein of the arm).
  Arms: Placebo (ZP8396)

SUMMARY:
The research study will investigate the safety and tolerability of ZP8396 in healthy study participants. In addition, the study will investigate how ZP8396 works in the body (pharmacokinetics and pharmacodynamics).

Participants will receive 1 single dose either as an injection under the skin (subcutaneous, s.c.) or an injection into a vein of one arm (intravenous, i.v.).

Participants will have 9 visits with the study team. One of these visits consists of 8 overnight stays at the study site. For each participant, the study will last up to 66 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Body Mass Index (BMI) between 21.0 and 29.9 kg/m^2, both inclusive
* Body weight of at least 70.0 kg
* Glycosylated hemoglobin A1c (HbA1c) less than 5.7 percent
* Further inclusion criteria apply

Exclusion Criteria:

* History of metabolic diseases more frequently associated with obesity, e.g. type-2-diabetes mellitus, hypertension, dyslipidemia, heart disease or stroke
* Systolic blood pressure < 90 mmHg or >139 mmHg and/or diastolic blood pressure less than 50 mmHg or greater than 89 mmHg
* Symptoms of arterial hypotension
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | From dosing (Day 1) to end of trial (Day 50)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ZP8396 (AUCτ) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Area under the plasma concentration-time curve over a dosing interval
Pharmacokinetics (PK) of ZP8396 (AUCinf) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics (PK) of ZP8396 (AUClast) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration
Pharmacokinetics (PK) of ZP8396 (Cmax) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Maximum (peak) plasma drug concentration
Pharmacokinetics (PK) of ZP8396 (tmax) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Time to reach maximum (peak) plasma concentration
Pharmacokinetics (PK) of ZP8396 (λz) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Elimination rate constant
Pharmacokinetics (PK) of ZP8396 (t½) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Elimination half-life
Pharmacokinetics (PK) of ZP8396 (Vz/f) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Apparent volume of distribution during terminal phase
Pharmacokinetics (PK) of ZP8396 (Vz) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Volume of distribution during the terminal phase (i.v. only)
Pharmacokinetics (PK) of ZP8396 (CL/f) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Apparent total clearance of the drug from plasma
Pharmacokinetics (PK) of ZP8396 (CL) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Total body clearance of the drug (i.v. only)
Pharmacokinetics (PK) of ZP8396 (MRT) | Day 1 (pre-dose) to Day 50 (1176 hours post-dose)
  Mean residence time
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (Cmax acetaminophen) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Maximum acetaminophen concentration after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (Tmax acetaminophen) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Time to maximum acetaminophen concentration after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (AUCacetaminophen, 0-60 min) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Area under the acetaminophen concentration-time curve from 0 to 60 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (AUCacetaminophen, 0-240 min) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Area under the acetaminophen concentration-time curve from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (Cmax, Plasma Glucose [PG]) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Maximum PG concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (Tmax, Plasma Glucose [PG]) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Time to maximum PG concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (AUCPG,0-60 min) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Area under the Plasma Glucose (PG) concentration-time curve from 0 to 60 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (AUCPG,0-240 min) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Area under the Plasma Glucose (PG) concentration-time curve from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (Cmax, insulin) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Maximum insulin concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (Tmax, insulin) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Time to maximum insulin concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (AUCinsulin,0-60 min) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Area under the insulin concentration-time curve from 0 to 60 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (AUCinsulin,0-240 min) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Area under the insulin concentration-time curve from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (Cmax, glucagon) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Maximum glucagon concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (Tmax, glucagon) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Time to maximum glucagon concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (AUCglucagon,0-60 min) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Area under the glucagon concentration-time curve from 0 to 60 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396, for dose cohorts greater than or equal to 0.7 mg (AUCglucagon,0-240 min) | 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 and Day 5
  Area under the glucagon concentration-time curve from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen

CONTACTS AND LOCATIONS:
Overall Officials: Zealand Pharma A/S, Study Director — Zealand Pharma A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No